CLINICAL TRIAL: NCT05782218
Title: HULA Study - Healthy Unique Lipids From Almonds
Brief Title: Healthy Unique Lipids From Almonds
Acronym: HULA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1950391; GH-22-DebedatJ-NR-01 (Other Grant/Funding Number: Almond Board of California)
Record Dates: First submitted 2023-02-17; First posted 2023-03-23 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-08

CONDITIONS: Nutrition, Healthy
Keywords: microbiome; cyclopropane; nutrition; unsaturated; fatty acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almond arm (Experimental): Almonds will be provided to increase the gut content in mono and poly-unsaturated fatty acids.
  Interventions: Dietary Supplement: Almonds
- Coconut arm (Experimental): This snack is isocaloric and almost perfectly matches the macronutrient profile of the almonds. However, despite being in the same quantity, almost all provided fatty acids will be saturated fatty acids.
  Interventions: Dietary Supplement: Coconut

INTERVENTIONS:
Dietary Supplement: Almonds — Participants will receive 2.2 oz (62 g) of almonds to ingest within 15 minutes.
  Arms: Almond arm
Dietary Supplement: Coconut — Participants will receive 1 oz (30 g) of a coconut-chocolate bar and 1.4 oz (40 g) of 100% dried coconut chips to ingest within 15 minutes.
  Arms: Coconut arm

SUMMARY:
This project will address the notion that "healthy" lipids such as monounsaturated fatty acids in almonds can be used by the bacteria living in our gut to generate "new" molecules with potentially interesting health properties. This metabolite pattern is anticipated to differ significantly when compared to non-almond foods rich in saturated fats.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 18 to 50 years of age
* Body mass index (BMI) categorized "normal" through "overweight" (18.5 - 29.9 kg/m2)
* Able to provide informed consent in English

Exclusion Criteria:

* pregnancy or lactation
* allergy or aversion to any of the foods that will be studied and/or provided
* history of gastrointestinal disorders including ulcerative colitis, Crohn's disease, celiac sprue, hereditary non-polyposis colorectal cancer (HNPCC), familial adenomatous polyposis, pancreatic disease, or liver disease
* history of metabolic diseases (type 2 diabetes, hyperlipidemia)
* previous gastrointestinal resection or bariatric surgery
* bleeding disorders that preclude blood draws
* recent hospital admissions (past 6 months) for heart disease (MI/CVA or CHF) or other CVD/CAD conditions under physician guided therapy that is not medically stable
* cancer under radiation or chemotherapy treatment that is active or within 6 months of treatment
* regular alcohol intake of > 2 drinks/day (equivalent to 720 mL of beer, 240 mL of wine, or 90 mL of spirits) and unwilling to abstain during the run-in week and test day
* use of tobacco and/or marijuana, hookahs, e-cigarettes (e-cigs, vapes, etc.) and not willing to abstain during the run-in week and test day
* use of illicit drugs and not willing to abstain during the run-in week and test day
* BMI ≥30 kg/m2
* regular (daily to weekly) use of over the counter (OTC) weight-loss aids, anti-acids or anti-inflammatories, and unwilling or unable to stop taking during the run-in week and test day
* regular OTC dietary supplements that interfere with the test foods being studied including pills, chewables, liquids or powders for the following: fiber, fish oil (including cod liver oil), probiotics, and unwilling or unable to stop taking during the run-in week and test day
* oral or IV antibiotic use in the past 6 months (could defer participation until 6 months post-completion of course of antibiotics)
* seated blood pressure >140/90 mmHg
* fasting clinical lab tests outside acceptable values as ascertained at the screening blood draw (Glucose (fasting), Urea, Creatinine, eGFR, Sodium, ALT/GPT, AST/GOT, Alk Phos, Total Bilirubin, Total protein, Albumin, Complete blood count, hematocrit, Total Cholesterol, HDL/LDL cholesterol, Triglycerides, Insulin Free, Total Insulin, Hemoglobin A1C)
* current use of specific prescription medication(s): Coumadin, Opiates within 1 month of study, Chlorthalidone, Canagliflozin, Tetracycline, Heparin, Anti-psychotics, Chlorothiazide, Dapagliflozin, Cephalosporin, Eliquis, Lithium, Hydrochlorothiazide, Empagliflozin, Penicillin, Indapamide, Insulin, Quinolone, Metolazone, Acarbose, Lincomycin, Oral Steroids within 1 month of study, Cholestyramine, Amiloride hydrochloride, Miglitol, Macrolide, RA / psoriasis medications, Colesevelam, Spironolactone, Liraglutide, Sulfonamide, Medications for rheumatologic / hematologic active disease, Colestipol, Triamterene, Metformin, Glycopeptide Abs, Ezetimibe, Furosemide, Aminoglycosides, Fenofibrate, Bumetanide, HIV/HAART therapy, Statins, Proton-pump inhibitors
* inability to freely give informed consent in English

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Change in the level of microbe-derived metabolites | One day (during the feeding day)
  Changes in the concentrations of microbe-derived metabolites in the blood and/or urine and/or stool of participants in the almond arm, versus a significantly different profile in participants in the coconut arm.

SECONDARY OUTCOMES:
Microbiome features associated with post-meal metabolite patterns | One day (during the feeding day)
  Positive or negative statistical associations between features in participants' gut microbiome and their post-meal changes in blood and/or urine and/or stool metabolites.

OTHER OUTCOMES:
Relationship between dietary habits and baseline (pre-meal) microbiota-derived blood metabolite levels in the baseline blood. | One day (inclusion visit)
  Positive or negative statistical associations between dietary habits and baseline circulating levels of microbial metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Debedat, PharmD/PhD, Principal Investigator — University of California, Davis; Sean H Adams, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No